CLINICAL TRIAL: NCT04412928
Title: Factors Affecting the Cure of Overactive Bladder Syndrome in Women Underwent Mid-urethral Sling Procedure
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Associate Professor, Far Eastern Memorial Hospital
Other Study IDs: 109048-E
Record Dates: First submitted 2020-05-31; First posted 2020-06-02 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mid-urethral sling procedure — mid-urethral sling procedure

SUMMARY:
We will estimate the incidence of patients with overactive bladder syndrome after surgery and explore related predictors.

DETAILED DESCRIPTION:
At present, around 30% of women with stress urinary incontinence have overactive bladder syndrome after mid-urethral sling procedure. But its predictive factor is still unclear. We will estimate the incidence of patients with overactive bladder syndrome after surgery and explore related predictors. In addition, we will explore the cure rate and predictors of cure of overactive bladder syndrome after the mid-urethral sling procedure for women with stress urinary incontinence. The above results will be used as a reference for preoperative and postoperative consultation.

ELIGIBILITY:
Inclusion Criteria:

* All women with stress urinary incontinence who underwent mid-urethral sling procedure from January 01, 2008 to July 31, 2019 will be reviewed.

Exclusion Criteria:

* Patients undergoing other gynecological operations at the same time, except for cystoscopy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with stress urinary incontinence
Study Population: All women with stress urinary incontinence who underwent mid-urethral sling procedure.
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Factors affecting the presence of overactive bladder syndrome after mid-urethral sling procedure | 10 year

SECONDARY OUTCOMES:
Factors affecting cure of overactive bladder syndrome after mid-urethral sling procedure | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No